CLINICAL TRIAL: NCT03710850
Title: Modification of Gut Microbiota in the Treatment of Insulin Resistance: a Personalized Approach
Acronym: TRIEMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Jan Gojda, MD, Head of unit, Charles University, Czech Republic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NV18-01-00040
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Insulin Resistance; Microbiome
Keywords: Insulin resistance; Diabetes; Inulin; Microbiome
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus | interventions — Inulin

STUDY DESIGN:
Intervention Model Description: single groups assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Responders (Experimental): Responders in terms of fecal butyrate production after acute inulin test.
  Interventions: Dietary Supplement: Inulin
- Non-responders (Experimental): Non-responders in terms of fecal butyrate production after acute inulin test.
  Interventions: Dietary Supplement: Inulin

INTERVENTIONS:
Dietary Supplement: Inulin — Inulin is a dietary fibre. Will be supplemented in a dose 10g/d for a period of 3 moths.

SUMMARY:
Gut microbiota may play a key role in many metabolic diseases, including type 2 diabetes (T2D). Consumption of high-fat/high-sugar western diet seem to alter human resident microbiota towards reduced genetic diversity and to influence its metabolic activity towards enhanced energy extraction. Plant-based diets are effective in the treatment of T2D but it is not clear whether their effect results solely from diet composition or whether it is mediated, at least partly, by different microbiota and its metabolic activity. One possible therapeutic approach is replacement of "pro-diabetic" microbiota with its "healthy" variant but what the "healthy" microbiota is and under which conditions this microbiota could stay stable and functional is not known. The aim of the proposed study is to identify possible metagenome/metabolome characteristics in different human cohorts (T2D vs vegans), to assess the stability of vegan microbiota in T2D-like environment and to evaluate the possibility to influence human T2D microbiota/metabolome towards more protective composition by dietary intervention.

DETAILED DESCRIPTION:
The aim of this project is to study the possibilities of gut microbiota manipulation in type 2 diabetes (T2D) towards more beneficial genetic and metabolic profile. This study address several issues. First, identification of specific metagenome/metabolome features characteristic for human cohorts with different risk of T2D development. Second, the resilience of microbiota associated with beneficial metabolic phenotype in pro-diabetogenic environment and the possibility to support its survival by prebiotic treatment. Third, development of the method for personalized prediction of the effectivity of prebiotic treatment in T2D patients and the evaluation of the benefit of long-term prebiotic administration in responders´ subpopulation. The project will be realized in three work packages.

WP1: Observation study focused on the description of gut microbiome and metabolome in obese type 2 diabetics, vegans and obese but otherwise healthy omnivores and identification of key markers specific for these populations.

WP2: Study focused on the interaction of vegan microbiota and pro-diabetogenic (western-type) diet and on the effects of prebiotic supplementation in germ-free animals. In addition, the effect of diet-alone and the effect of standardized Schaedler flora will be tested as well.

WP3: The identification of predictive markers indicative for the benefit of prebiotic treatment in the individual context (T2D cohort) and second, long-term human intervention study in the selected responders´ group aimed on the possibility of therapeutic modulation of gut microbiome/ metabolome by prebiotics. Only WP3 is subjected to clinical trial registration.

In details:

WP 3: Identification of T2D subpopulations according to their susceptibility to dietary fiber intervention Questions:

1. Are there different subpopulations within T2D subjects that differ in their ability to increase SCFA production in response to prebiotic supplementation?
2. Is it possible to identify these subpopulations ("responders" vs "non-responders") by simple intervention test?
3. Is this phenomenon associated with specific microbiota composition?
4. Within "responder" subpopulation, is it possible to manipulate fecal metabolome/metagenome towards more beneficial composition by long-term prebiotic intervention? In order to fulfill this task microbiome characterization of T2D cohort in WP1 will be used.

The aim of WP3 is to provide the proof of concept that a diet enriched with specific prebiotics improves the specific (SCFA) metabolite production and that the beneficial effect is dependent on pre-existing microbiota composition.

Acute intervention test ("inulin test") The participants enrolled into T2D cohort will be asked to participate in short-term intervention test. They will be provided the prebiotic and instructed on the test procedure.

Step 1: sample the stool ("sample 1"); step 2: take the dose (20 g) of inulin; step 3: during following three days collect sample of feces at each defecation. The samples will be analyzed by NMR and mass spectrometry with special respect to SCFA content.

Primary readout: The magnitude of SCFA content elevation after the bolus prebiotic administration.

Secondary readout: The potential association between the response to prebiotic bolus and microbiota composition.

Long-term intervention study Based on the results of acute inulin intervention test, the subgroups of most pronounced "responders" and "non-responders" will be selected (defined as both extreme tertiles of the group, at least 10 subjects are expected to be enrolled per subgroup). Participants from both subgroups will be asked to take part in three months intervention study when they will be administered 10 g of inulin prebiotic (FAN s.r.o., Tišice 225, 27715 Tišice) on every-day basis. Prior and at the end of the intervention period, the participants will be subjected to metabolic characterization, indirect calorimetry and assessment of intestine permeability. Feces samples will be collected before the study and then after each month for 16S rRNA sequencing, NMR spectroscopy and mass spectrometry.

Primary readout:

gut microbiome and fecal, urine and plasma metabolome composition of feces

Secondary readouts:

1. metabolic characteristics: basal blood tests (glucose, lipid profile, NEFA, insulin, C-peptide); twostep hyperinsulinemic euglycemic clamp; indirect calorimetry with energy expenditure and respiratory quotient
2. intestinal permeability markers: serum content of bacterial endotoxin, D-lactate, endotoxin core antibody, iFABP and citrulline.

Expected outcome: validation of short prebiotic intervention test as a tool for prediction of the efficiency and benefit of long-term prebiotic supplementation; evaluation of the benefit of long-term prebiotic supplementation in T2D "responder" subgroup.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese volunteers (BMI over 25)

Exclusion Criteria:

* diabetes on medication
* any disease known to affect intestinal permeability
* antibiotic use less than 3 months prior to enrollment
* gravidity/lactation in women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Butyrate production | 3 months
  Fecal butyrate content
Glucose disposal | 3 months
  Rate of glucose disposal from 80IU insulin glucose clamp

SECONDARY OUTCOMES:
Suppression of lipolysis | 3 months
  Decrease in plasma levels of glycerol/NEFA in 10IU insulin glucose clamp

CONTACTS AND LOCATIONS:
Overall Officials: Jan Gojda, MD, PhD, Principal Investigator — Charles University, Czech Republic
Locations (1):
- University Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No